CLINICAL TRIAL: NCT06248359
Title: Association Between Early Postoperative L-Arginine Administration and Acute Kidney Injury Following Cardiac Surgery
Brief Title: Association Between Postoperative Administration of L-Arginine and CSA-AKI
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Other Study IDs: KY20232170-C-1
Record Dates: First submitted 2024-01-24; First posted 2024-02-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arginine Use: At least one dose of L-arginie was administered in the early postoperative stage
  Interventions: Drug: L-Arginine hydrochloride
- Without Arginine: No L-arginie was administered

INTERVENTIONS:
Drug: L-Arginine hydrochloride — Postoperative administration of L-Arginine hydrochloride before incidence of CS-AKI
  Groups: Arginine Use

SUMMARY:
To investigate the association between the the early administration of L-Arginine after CPB-assisted cardiac surgery and the incidence of CS-AKI in adult patients. To test if it can reduce the incidence of post-operative AKI.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (over 18 years)
* underwent CPB assisted cardiac surgery
* admitted to ICU

Exclusion Criteria:

* congenital heart disease
* underwent deep hypothermic circulatory arrest (DHCA)
* with glomerular filtration rate (eGFR) below 30 mL/min/1.73 m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were admitted to the ICU after cardiac surgery with CPB.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative AKI | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 30 days
  Serum Creatinine Criteria:
  Increase in Serum Creatinine:
  An absolute increase in serum creatinine of 0.3 mg/dL (26.5 µmol/L) within 48 hours.
  OR a percentage increase in serum creatinine of ≥50% within 7 days. These criteria are relative to the baseline creatinine level, which is usually the recent preadmission value.
  Urine Output Criteria:
  Oliguria, defined as a urine output <0.5 mL/kg/h for more than 6 hours. OR anuria, defined as a urine output <100 mL in 24 hours.

SECONDARY OUTCOMES:
Renal failure | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 30 days
  KDIGO defined AKI stage ≥ 2, or if dialysis is required for newly developed conditions
  KDIGO classifies AKI into three stages based on the severity:
  Stage 2:
  Increase in serum creatinine of 2.0 to 2.9 times baseline OR Urine output <0.5 mL/kg/h for ≥12 hours.
  Stage 3:
  Increase in serum creatinine of 3.0 times baseline OR Increase in serum creatinine to ≥4.0 mg/dL OR Initiation of renal replacement therapy (RRT) OR Urine output <0.3 mL/kg/h for ≥24 hours OR anuria for ≥12 hours.
in-hospital mortality | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 30 days
  all-cause postoperative deaths observed
length of in-hospital stay | from the time of end of surgery until time of documented hospital discharge or time of death, whichever came first, assessed up to 30 days
  postoperative stay until discharge or death

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No